CLINICAL TRIAL: NCT02562196
Title: Effect of Transcranial Direct Current Stimulation (tDCS) Optimized Protocol for the Treatment of Migraine
Brief Title: tDCS for the Treatment of Migraine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Effect of Transcranial Direct Current Stimulation (tDCS) Optimized Protocol for the Treatment of Migraine, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Effect_tDCS_Migraine
Record Dates: First submitted 2015-09-22; First posted 2015-09-29 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Migraine Disorders
Keywords: migraine disorders; transcranial direct current stimulation; electric stimulation therapy; pain
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- optimized protocol chosen (Experimental): a randomized, sham-controlled, double-blinded and parallel group trial (12 therapeutic sessions) with optimal protocol (defined in phase 1) and sham tDCS will be conducted to evaluated electrical cortical activity and pain control, number of migraine attacks and quality of life of migraine patients. An interval of 48hs between sessions will be taken.
  Interventions: Device: tdcs
- sham tDCS (Sham Comparator): a randomized, sham-controlled, double-blinded and parallel group trial (12 therapeutic sessions) with optimal protocol (defined in phase 1) and sham tDCS will be conducted to evaluated electrical cortical activity and pain control, number of migraine attacks and quality of life of migraine patients. An interval of 48hs between sessions will be taken.
  Interventions: Device: tdcs

INTERVENTIONS:
Device: tdcs — The direct electric current will be applied by surface electrodes with 35cm² and composed of rubbers conductive electricity and surrounded by sponges soaked in saline solution. The electrodes position will be performed according the 10-20 international system of marking and the different montages will be realized by distinct applications sites.
  To stimuli the primary motor cortex the active electrode will be positioned on C3 point and the reference electrode on the contralateral supraorbital region. To visual cortex stimulation, the active electrode will be positioned on the Oz point and the reference on Cz. To duo stimulation, the two electrodes will be considerate actives, stimulating the visual and motor cortex simultaneously. The sham tDCS has already been used in several studies to assess the effect active tDCS and the duration of the current is only 30 seconds.

SUMMARY:
The aim of this study is to evaluate an optimized protocol of tDCS that normalize the lack of habituation and efficiency of inhibitory cortical circuits in migraine patients. For this purpose, migraineurs volunteers will undergo to optimized tDCS protocol or sham tDCS.

DETAILED DESCRIPTION:
A randomized, sham-controlled, double-blinded and parallel group trial (12 therapeutic sessions) with optimal protocol (defined in phase 1) and sham tDCS will be conducted to evaluated electrical cortical activity and pain control, number of migraine attacks and quality of life of migraine patients. Electrical cortical activity will be assessed through: (i) motor evoked potential (MEP); (ii) motor threshold (MT); (iii) short interval intracortical inhibition (SICI); (iv) intracortical facilitation (ICF); (v) phosphene threshold (PT) and (vi) visual evoked-potential (VEP-habituation). Clinical outcomes will be evaluated through: (i) headache diary; (ii) visual analog scale (VAS); (iii) Migrainde disability assessment (MIDAS); (iv) Headache Impact Test (HIT-6) and (v) World Health Organization quality of life assessment instrument (WHOQOL BREF).

ELIGIBILITY:
Inclusion Criteria:

* Presented diagnostic of episodic migraine with or without aura or probably migraine with or without aura according to the criteria for diagnosis of International Classification of Headache Disorders (ICHD-III)
* Disease duration of at least 12 months
* Without preventive medication for at least 6 months prior to initiation of treatment

Exclusion Criteria:

* Pregnant women;
* Pacemaker;
* History of seizures;
* Metallic implants in the head;
* Patients with clinical evidence of brain injuries;
* Chronic pain associated to others diseases;
* Use of neuroleptic medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-08 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change in headache diary variables | 3 followed months
  it will be evaluated the number of migraine attacks, pain intensity, duration of each attack and number of painkillers intake. Patients will answer this diary during all experimental period (months).

SECONDARY OUTCOMES:
Changes on Visual Evoked Potentials measures | at baseline, 1 month and 2 months, 3 months
  volunteers will be invited to sit in a comfortable chair, in a calm and dark room, at 90 cm of distance from computer screen. It will be asked to fix his right eye visual field on a red point at the center of the screen (the left one will be blindfolded). Visual stimuli will be a black and White grid pattern, alternating at a frequency of 3.1 Hz. Electrodes used to record data will be localized on Oz and Fz points according International 10-20 system. During the test, 600 cortical answers will be recorded. Data will be collected and recorded in a personal computer, and after, converted to the ".txt" format to futures analysis with MATLAB.
Changes on HIT-6 | at baseline, 1 month and 2 months, 3 months.
  this is a questionnaire, composed of six questions, developed to measure the impact of headache on daily living activities of individuals with chronic episodic and migraine. It is a valid and reliable instrument for this population and its results are related to clinic parameters of migraine, e.g. severity and quality of life. Total score ranges from 36 to 78 and it is categorized into four levels: slight or no impact (38 to 49 points); some impact (50 to 55 points); substantial impact (56-59 points); very severe impact (60 or more points). The minimum important difference for this scale was estimated at -2.5 to -5.5 points (within groups) and -1.5 points (between groups).
Changes on MIDAS | at baseline, 1 month and 2 months, 3 months.
  this is a questionnaire, composed of five items, created to evaluate disability caused by headache in a period of 3 months. This instrument is reliable and validated in several countries, and its Portuguese version may be used to identify severe cases of migraine. MIDAS total score will be obtained by adding days lost in each of the areas being categorized into four levels: slight or none disability (0 to 5 days); mild disability (6 to 10 days); moderate disability (11 to 20 days); intense capacity (≥21 days).
Changes on VAS | at baseline, 1 month and 2 months, 3 months.
  this scale will be used to measure the patients' pain intensity. VAS is an important instrument to verify, reliably, the patient's evolution during treatment. This scale will be used at beginning and end of each period (observation and treatment), before and after each tDCS session. For the VAS use, pain intensity will be asked to the patient. 0 cm means total pain absence and 10 cm is the level of maximum pain bearable by the patient.
Changes on motor evoked potentials | through study completion, assessed up to 1 month (before and after each section)
  to measure MEP, the intensity of the magnetic stimulator will be adjusted to 120% of rest motor threshold and 10 stimuli will be registered. For evaluation volunteers will be instructed to sit in a chair and get into a comfortable position. Initially, single-pulse transcranial magnetic stimulation (TMS) will be administered over the motor cortex to determine the cortical representation area of the first dorsal interosseous muscle (FDI). For all evaluations the same figure-eight coil is used, in order to avoid measurement bias. Amplitude means of evoked potentials will determine the MEP.
Changes on inhibition and facilitation | through study completion, assessed up to 1 month (before and after each section)
  to evaluate these variables, subthreshold conditioning stimuli (80% of RMT) and suprathreshold test stimuli (120% of RMT) will be delivered at an inter stimulus intervals (ISI) of 2 milliseconds, to determine the short interval cortical inhibition (SICI). The Intracortical facilitation (ICF) will be evaluated by the MEP average at an ISI of 10 milliseconds. Ten stimulus will be applied in each condition (unconditioned pulse, and pairs of stimuli with ISI of 2 and 10 milliseconds). The order of stimulus delivered will be pseudorandomized and SICI and ICF will be expressed as a percentage of a conditioned stimuli in regarding an unconditioned stimuli.
Changes from phosphene threshold | through study completion, assessed up to 1 month (before and after each section)
  a 10-cm circular coil was used that has giving a peak magnetic field strength of 2 tesla. Subjects were asked to wear a blindfold, sit comfortably in a chair and to close their eyes to diminish ambient light.In sagittal line, three points were scored: 2, 3 and 4 cm above the inion. The single pulse TMS was applied to one of the points scored and the subject was asked to report the presence or absence of a phosphene immediately after stimulation. The stimulation was repeated ten times at each intensity with a maximum frequency of 0.2 Hz, stimulation was initially applied to 60% of the maximum intensity of the stimulator. The intensity of stimulation was changed into blocks of 5% to minimum intensity that the subject can perceive the phosphene certainly, five times ten, then this value was set as the PT.

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Monte-Silva, PhD, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil